CLINICAL TRIAL: NCT05616741
Title: A Randomized, Wait-list Controlled Trial of Daily, Home-based Biofeedback Therapy Using Cerebri for the Prevention of Migraine Attacks in Adults With Episodic Migraine
Brief Title: Home-based Biofeedback for the Prevention of Migraine
Acronym: BioCer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordic Brain Tech AS (Other Government)
Collaborators: Norwegian University of Science and Technology (Other); St. Olavs Hospital (Other); University Hospital, Akershus (Other); Haukeland University Hospital (Other); University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 502734; CIV-NO-22-08-040446 (Other: EUDAMED)
Record Dates: First submitted 2022-10-25; First posted 2022-11-15 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: This study is an open-label, randomized, wait-list controlled multicenter trial with a run-in phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Cerebri biofeedback and Cerebri headache diary
  Interventions: Device: Cerebri biofeedback; Other: Cerebri headache diary
- Waitlist control group (Other): Only Cerebri headache diary
  Interventions: Other: Cerebri headache diary

INTERVENTIONS:
Device: Cerebri biofeedback — Daily use of a mobile application connected with two wireless sensors for measurement of muscle tension, heart rate variability, and peripheral finger temperature, to be used for home-based biofeedback treatment.
  Arms: Treatment group
Other: Cerebri headache diary — Daily registration of headache and medication with the Cerebri mobile application. This intervention is identical for both study arms.

SUMMARY:
The goal of this clinical trial is to test an app-based biofeedback treatment in adults with migraine. The aim of the study is to investigate the safety and effectiveness of biofeedback treatment using the medical device Cerebri, compared to wait-list controls.

Participants will perform 10 minutes biofeedback daily, in addition to daily registrations in the headache diary. Wait-list controls will complete daily registrations in the headache diary during the same period.

Researchers will compare the reduction in the number of days with migraine from baseline per 28-day period between treatment group and the wait-list group.

DETAILED DESCRIPTION:
This trial, BioCer, is a clinical study to test the effectiveness and safety of the app-based biofeedback treatment, Cerebri, for migraines in adults. Bodily signals that are thought to be associated with migraines are measured by sensors during biofeedback. During the treatment, one sensor is attached to the shoulder to measure activity in the shoulder and neck muscles and one sensor is attached to the index finger to measure temperature and heart rate variability. By getting on-screen feedback on the phone, the user can learn techniques to reduce muscle tension, and increase finger temperature and heart rate variability. Reduced muscle tension, as well as an increase in finger temperature and heart rate variability is a sign of relaxation and a deactivation of the nervous system, which can lead to fewer and less serious migraine attacks. The aim of the study is to investigate the safety and effectiveness of biofeedback treatment using Cerebri compared to wait-list controls.

In this study, the investigators will recruit 286 adults with episodic migraines. All participants will complete one month of daily headache diary entries in the Cerebri app without any specific treatment. This will serve as the "baseline" measurements. Subsequently, the participants will be randomized to either the treatment group or the wait-list group. The treatment group will conduct daily biofeedback sessions of 10 minutes duration for 12 weeks. The wait-list group does not receive any specific treatment for 12 weeks but serves as an important basis for comparison to evaluate the treatment effect. The wait-list control group will be offered active treatment for 12 weeks after the initial 12-week wait-list period is completed. Participants in both groups (the treatment group and the wait-list control group) must complete daily registrations in the headache diary included in the app.

The primary endpoint of the study is the change in the number of days with migraine per 28-day period. The reduction in the number of migraine days will be compared between the treatment group and the wait-list group. Secondary endpoints include the change in intensity of headaches, the change in consumption of acute medication for migraine, and the number of participants with at least a 30% reduction in the number of migraine days.

There is a wide range of preventive treatments for migraines, both drug and non-drug, but many have limited effects and potentially numerous side effects. If the biofeedback app proves to be effective, it may represent a useful and viable treatment option for episodic migraine patients, that is readily available and unlikely to cause unwanted side effects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age inclusive or older, at the time of signing the informed consent
* Episodic migraines with or without aura diagnosed by a neurologist/physician per International Classification of Headache Disorders 3rd edition (ICHD-3).
* History of at least 4 and up to 14 days of migraines per 28-day period in the 3 months prior to screening (as recalled by the subject). This frequency must be confirmed in the headache diary before randomization to treatment or wait-list control.
* At least three months of experience with smartphone and access to an iOS or Android phone at home.
* Capable of giving signed informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Onset of migraine before age 50 years.

Exclusion Criteria:

* More than 14 days of headache (all types) per 28-day period.
* Subjects diagnosed with trigeminal autonomic cephalalgias and neuralgias.
* Subjects with secondary headache conditions.
* Subject with pathologies that inhibit use of the device according to the instructions for use (e.g., blindness, deafness).
* Use of non-pharmacological preventive treatment (meditation, physical therapy, psychotherapy as a headache treatment, acupuncture, etc.), with the exception of stable treatment for other indications than migraine
* Use of concurrent migraine preventive medication, with the exception of stable dose (≥3 months) monotherapy of migraine preventive medication · Subjects who have previously attempted three or more prophylactic pharmacological treatments in adequate doses, without significant clinical effect.
* Subjects taking opioids (>3 days per month) or barbiturates at the time of screening.
* Subject participates in another clinical investigation or has participated in CER-MIG-1.
* Alcohol overuse or illicit drug use.
* Subject who is unlikely to follow Clinical Investigation Plan or where treatment seems futile in the opinion of the Investigator or have demonstrated an inability to sufficiently adhere to headache diary entries (<70%).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Efficacy of intervention in treatment group compared to the wait-list control group in reducing the frequency of migraine days | 4 months
  Change in the mean number of migraine days from baseline to the last 28-day period during the treatment phase, in the treatment group as compared to the wait-list control group

SECONDARY OUTCOMES:
Early onset efficacy of intervention in treatment group compared to the wait-list control group in reducing the frequency of migraine days | 4 months
  Change in the mean number of migraine days from baseline to the first two 28-day periods during the treatment phase, in the treatment group as compared to the wait-list control group
Efficacy of intervention in treatment group compared to the wait-list control group in reducing migraine intensity | 4 months
  Change in the mean intensity of migraine/headache using 11-point scale (0-10), where high score means high migraine intensity. Change will be assessed from baseline to the last 28-day period during the treatment phase, in the treatment group as compared to the wait-list control group
Proportion of participants with at least 30% reduction in migraine days between the treatment and wait-list control groups | 4 months
  Responder rate, defined as the number of participants with at least a 30% reduction in migraine days from baseline to the last 28-day period, in the treatment group as compared to the wait-list control group.
Change in acute migraine drug use between the treatment and wait-list control groups | 4 months
  Change in acute migraine drug treatment use from baseline to the last 28-day period, in the treatment group as compared to the wait-list control group.
Change in subject-reported headache-related disability from baseline to treatment between the treatment and control groups | 4 months
  Change in subject-reported headache-related disability measured by Migraine-Specific Quality of Life Questionnaire version 2.1 (MSQ v2.1) from baseline to the last 28-day period, in the treatment group as compared to the wait-list control group. The MSQ v2.1 contains 14 questions from three domains with six response alternatives ranging from "none of the time" to "all of the time". Low score indicates low amount of headache-related disability.

OTHER OUTCOMES:
Change in weekly migraine days during the treatment period (for trend analyses) | 4 months
  Description of change from baseline in weekly migraine days in treatment group.
Change in 28-day period headache days | 4 months
  Change from baseline in the mean number of headache days for each 28-day period in treatment group.
Adherence to protocol | 4 months
  A description of subjects' adherence to the protocol in treatment group assessed by proportion of completed biofeedback sessions and proportion of completed headache diary entries.
Adherence to the headache diary in the Cerebri mobile application | 4 months
  A description of the frequency of headache diary entries in the Cerebri mobile application in the treatment group.
Change in the patient's impression of overall health | 4 months
  Mean self-reported Patient Global Impression of Change (PGI-C) score in treatment group. Possible scores range from 1 to 7, where 1 indicates positive change, 7 indicates negative change and 4 is neutral.
Change in frequency of migraine days during add-on treatment period in wait-list control group | 7 months
  Change from baseline and wait-list period in the mean number of migraine days for each 28-day period during the add-on treatment period in the wait-list group.
To describe any treatment-emergent adverse events encountered during the investigation | 4 months
  A description of the frequency and severity of treatment-emergent adverse events, ADEs, SADEs, and USADEs).

CONTACTS AND LOCATIONS:
Overall Officials: Tore Meisingset, MD, PhD, Principal Investigator — St. Olavs Hospital
Locations (4):
- Norway (4):
  - Akershus University Hospital HF, Lørenskog, Akershus
  - Haukeland University Hospital HF, Bergen
  - University Hospital of North Norway, Tromsø
  - St.Olavs Hospital HF, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poole AC, Stubberud A, Simpson M, Oie L, Skalstad ETV, Bjork MH, Kristoffersen ES, Vetvik KG, Olsen A, Larsen ICK, Linde M, Tronvik EA, Meisingset TW. Biofeedback therapy using Cerebri for the prevention of migraine attacks in adults with episodic migraine (BioCer): a randomized, wait-list controlled trial - the study protocol. F1000Res. 2025 Aug 29;13:775. doi: 10.12688/f1000research.149807.2. eCollection 2024. PMID 40909914